CLINICAL TRIAL: NCT04157452
Title: Prediction of Sepsis After Flexible Ureteroscopy in Patients With Proximal Ureteral Stone by Using Preoperative Factors
Brief Title: Prediction of Sepsis After Flexible Ureteroscopy
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Li Cong, Professor, Tongji Hospital
Other Study IDs: 2019S1035
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Urolithiasis; Sepsis; Surgery--Complications
MeSH Terms: conditions — Urolithiasis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- proximal ureteral stone patient
  Interventions: Procedure: flexible ureteroscopy

INTERVENTIONS:
Procedure: flexible ureteroscopy — flexible ureteroscopy is used to removed the stone. If a double-J stent was inserted pre-operatively, it was removed at the beginning of surgery. Rigid ureteroscopy was routinely used for ureteral dilatation before fURS. A 0.035 mm guidewire was advanced through the urethral and ureteral meatuses to the renal pelvis under direct rigid ureteroscope vision. A 14-Fr ureteral access sheath (Cook Medical, Bloomington, IN) was then passed over the wire to the ureteropelvic junction, and 7.5-Fr fURS (Flex-X2, Karl Storz, Germany) was performed through the sheath. Intrarenal pressure was stabilized by a pressure-sensitive pump (Shenda Medical, China). Holmium: yttrium-aluminum-garnet laser was used to fragment the stones. After lithotripsy, 6-Fr double-J stent was routinely inserted in all cases for 2-4 weeks.

SUMMARY:
Sepsis is a lethal complication of flexible ureteroscopy. The aim of this study is to identify predictors of sepsis after flexible ureteroscopy in patients with solitary proximal ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

* history of fURS to treat unilateral, solitary, and proximal ureteral stones
* age ≥18 years

Exclusion Criteria:

* anatomical renal abnormalities such as transplant kidney, solitary kidney, horseshoe kidney, and kidney duplication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are enrolled in Wuhan Tongji Hospital from January 2012 to December 2018. Patient data is collected from institutional medical record archives.
Sampling Method: Non-Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
complication-sepsis | within 48 hour after surgery
  sepsis is defined as the concurrence of infection and at least 2 of the following 4 criteria: (1) body temperature >38°C, (2) heart rate >90/minute, (3) respiratory rate >20/minute, and (4) leukocyte count <4,000 cells/μL or >12,000 cells/μL

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China